CLINICAL TRIAL: NCT01080885
Title: Linking Home Environments and Primary Care: Obesity Prevention for 2-5 Year Olds
Brief Title: Healthy Homes/Healthy Kids Preschool
Acronym: HHHK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 08-149; R21DK078239-01A2 (NIH)
Record Dates: First submitted 2010-03-03; First posted 2010-03-04 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2012-04

CONDITIONS: Obesity
Keywords: Prevention; Prevention of unhealthy weight gain
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Busy Bodies/Better Bites (Experimental): Healthy Eating/Physical Activity Intervention
  Interventions: Behavioral: Busy Bodies/Better Bites
- Healthy Spots/Safe Tots (Active Comparator): Injury Prevention and Safety Intervention
  Interventions: Behavioral: Healthy Spots/Safe Tots

INTERVENTIONS:
Behavioral: Busy Bodies/Better Bites — This intervention will include brief counseling from the pediatrician paired with a 6 month home-based program delivered via phone by a masters-level health behavior specialist to promote implementation of the healthy eating and physical activity home environmental strategies.
  Arms: Busy Bodies/Better Bites
Behavioral: Healthy Spots/Safe Tots — This intervention will include the same brief counseling from the pediatrician paired with a 6 month home-based program delivered via phone by a masters-level health behavior specialist to promote implementation of the safety and injury prevention home environmental strategies.
  Arms: Healthy Spots/Safe Tots

SUMMARY:
The goals of this study are to evaluate the feasibility, acceptability, and potential efficacy of an innovative obesity prevention intervention integrating pediatrician counseling and a home-based program to prevent unhealthy weight gain among 2-4 year old children at risk for obesity.

DETAILED DESCRIPTION:
The pediatric primary care setting is a relatively untapped resource for addressing obesity prevention. The goals of this developmental study are to develop and evaluate the feasibility and acceptability of a primary care-based, preschool obesity prevention intervention integrating pediatrician counseling and a home-based program for parents of 2-4 year old children at risk for obesity. We propose to recruit 60 parent-child dyads from families of 2-4 year old at risk children (e.g., BMI between the 85th and 95th percentile for age and gender or a BMI between the 50th and 85th percentile and at least one overweight parent) and randomize each dyad to one of the following groups: (a) Healthy Eating/Physical Activity Intervention including brief pediatrician counseling regarding the child's current BMI%ile status, recommendations for home environmental changes to achieve a healthy weight gain trajectory, and home safety and injury risk reduction recommendations paired with a 6 month home-based program delivered via phone by a health behavior specialist to promote implementation of the obesity prevention home environmental strategies, or (b) General Health/Safety/Injury Prevention Contact Control Intervention: Families will receive the same brief counseling from their pediatrician paired with a 6 month home-based program delivered via phone by a health behavior specialist to promote implementation of the general health, safety and injury prevention home environmental strategies.

* Healthy Eating/Physical Activity Home-based Intervention: The "Busy Bodies/Better Bites" intervention arm will include brief pediatrician counseling regarding the child's current BMI percentile status, recommendations for home environmental changes to achieve a healthy weight gain trajectory, and home safety and injury risk reduction environmental recommendations paired with a 6 month home-based program delivered via phone by a masters-level health behavior specialist to promote implementation of the obesity prevention home environmental strategies.
* Safety/Injury Prevention Home-based Contact Control Intervention: The "Healthy Tots/Safe Spots" intervention arm will include the same brief counseling from the pediatrician paired with a 6 month home-based program delivered via phone by a masters-level health behavior specialist to promote implementation of the safety and injury prevention home environmental strategies.

ELIGIBILITY:
Inclusion Criteria:

1. BMI between the 85th and 95th percentile for age and gender or
2. BMI between the 50th and 85th percentile and at least one overweight parent (BMI ≥ 25 kg/m2)
3. Receives care at a HealthPartners Clinic in the Twin Cities Metropolitan Area

Exclusion Criteria:

1. Children with the following chronic conditions: kidney disease, Type 1 diabetes, lupus, a thyroid condition, cancer or a chromosomal abnormality such as Down's syndrome or Turner's syndrome.
2. Children who within the last six months or who those who are currently taking the following medications and took them or will be taking them for more than a month: Prednisone, Prednisolone and Decadron.
3. Families who have limited English skills.
4. Families who plan to move out of the metropolitan area within the next six months.

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2010-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Parent and pediatrician participation and satisfaction | 6 months
  Parents of at risk preschool children and pediatricians will show high participation rates in and report high levels of satisfaction with the interventions.
Healthy Eating | 6 months
  Healthy Eating/Physical Activity Home-based Intervention participants will show lower levels of sweetened beverage and higher levels of lower fat/calorie snack and meal consumption compared to Safety/Injury Prevention Home-based Contact Control Intervention participants. The Nutrition Data System for Research will be used to measure this change.
Levels of TV watching | 6 months
  Healthy Eating/Physical Activity Home-based Intervention participants will show lower levels of TV watching compared to Safety/Injury Prevention Home-based Contact Control Intervention participants;
Physical activity levels | 6 months
  Healthy Eating/Physical Activity Home-based Intervention participants will show higher levels of physical activity compared to Safety/Injury Prevention Home-based Contact Control Intervention participants. Physical activity level will be measured by accelerometry.

SECONDARY OUTCOMES:
Hypothesized mediators of BMI change | 6 months
  Parents in the Healthy Eating/Physical Activity Home-based Intervention will report more favorable levels of hypothesized mediators of BMI change (e.g., family meal frequency, availability of lower fat/calorie foods and physical activity opportunities) compared to Safety/Injury Prevention Home-based Contact Control Intervention participants.
Body mass index (BMI) percentile | 6 months
  Participation in the Healthy Eating/Physical Activity Home-based Intervention will lead to reduced BMI percentile compared to Safety/Injury Prevention Home-based Contact Control Intervention participant.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy E Sherwood, PhD, Principal Investigator — HealthPartners Institute
Locations (1):
- HealthPartners Research Foundation, Bloomington, Minnesota, United States